CLINICAL TRIAL: NCT07324044
Title: Chrono-ALIGN Trial: The Impact of Chronotype-Based Chrono-Nutrition on Metabolic Health, Gut Microbiota, Appetite, and Circadian Alignment in Post-Bariatric Surgery Patients: A Randomized Controlled Trial
Brief Title: Chrono-ALIGN: A Chronotype-Based Chrono-Nutrition Intervention in Post-Bariatric Patients
Acronym: Chrono-ALIGN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Amani Al-Farraj, Ms., King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chrono-ALIGN
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Obesity (Disorder); Morbid Obesity; Bariatric Sleeve Gastrectomy; Meal Time; Chronotype; Circadian Rhythm
Keywords: chrononutrition; Bariatric Surgery; Gastric Sleeve; Gut Microbiota; Appetite; Meal Timing
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design with three arms. Participants will be randomized in a 1:1:1 ratio to (1) standard post-bariatric nutritional care without specific meal timing (Control), (2) early time-restricted eating (eTRE); or (3) chronotype-based chrono-nutrition (CB-CN; meal timing tailored to individual chronotype using the Munich Chronotype Questionnaire). Each intervention follows bariatric guidelines emphasizing protein adequacy, hydration, and micronutrient supplementation. The model is designed to evaluate whether aligning meal timing with chronotype improves weight loss maintenance, metabolic health, gut microbiota composition, epigenetic regulation, and psychological outcomes at 12 months
Who Masked: Outcomes Assessor
Masking Description: Due to the behavioral nature of the dietary interventions, participants and care providers cannot be blinded. However, outcome assessors, including laboratory personnel and data analysts, will remain blinded to group allocation to minimize detection and analysis bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Post-Bariatric Care (Active Comparator): Participants receive routine post-bariatric nutritional care with no prescribed meal-timing window. Dietitians provide standard guidance on protein adequacy (~60-80 g/day unless otherwise indicated), hydration, and routine micronutrient supplementation per clinic practice. Follow-ups occur at 3, 6, and 12 months; outcomes include body weight, metabolic markers, appetite-related hormones, questionnaires, wearables, and stool samples. This arm controls for the effects of usual care and non-timing dietary counseling.
  Interventions: Behavioral: Standard Post-Bariatric Care (Control)
- Early Time-Restricted Eating (eTRE) (Experimental): Participants consume all caloric intake within a fixed daytime 10-hour window (08:00-18:00) on ≥6 days/week. Water/unsweetened tea/black coffee are allowed outside the window. Diet composition follows bariatric guidelines (protein ~60-80 g/day, hydration, routine micronutrients). Dietitians provide structured meal-timing plans and problem-solving support; timing logs and wearables document adherence. Assessments at 3, 6, and 12 months mirror the control arm.
  Interventions: Behavioral: Early Time-Restricted Eating (eTRE)
- Chronotype-Based Chrono-Nutrition (CB-CN) (Experimental): Meal timing is personalized to chronotype (morning/intermediate/evening) determined with the Munich Chronotype Questionnaire (MCTQ). Plans target an earlier first meal and completion of the last meal ≥3-4 h before habitual bedtime, with an eating window of ~10 h/day on ≥6 days/week, adjusted to chronotype using stepwise phase-advance strategies where needed. Diet composition follows bariatric guidelines (protein, hydration, micronutrients). Timing logs and wearables track adherence; visits at 3, 6, and 12 months.
  Interventions: Behavioral: Chronotype-Based Chrono-Nutrition (CB-CN)

INTERVENTIONS:
Behavioral: Standard Post-Bariatric Care (Control) — Participants receive routine post-bariatric nutritional care with no prescribed meal-timing window. Dietitians provide standard guidance on protein adequacy (~60-80 g/day unless otherwise indicated), hydration, and routine micronutrient supplementation per clinic practice. Follow-ups occur at 3, 6, and 12 months; outcomes include body weight, metabolic markers, appetite-related hormones, questionnaires, wearables, and stool samples. This arm controls for the effects of usual care and non-timing dietary counseling.
  Arms: Standard Post-Bariatric Care
Behavioral: Early Time-Restricted Eating (eTRE) — Participants consume all caloric intake within a fixed daytime 10-hour window (08:00-18:00) on ≥6 days/week. Water/unsweetened tea/black coffee are allowed outside the window. Diet composition follows bariatric guidelines (protein ~60-80 g/day, hydration, routine micronutrients). Dietitians provide structured meal-timing plans and problem-solving support; timing logs and wearables document adherence. Assessments at 3, 6, and 12 months mirror the control arm.
  Arms: Early Time-Restricted Eating (eTRE)
Behavioral: Chronotype-Based Chrono-Nutrition (CB-CN) — Meal timing is personalized to chronotype (morning/intermediate/evening) determined with the Munich Chronotype Questionnaire (MCTQ). Plans target an earlier first meal and completion of the last meal ≥3-4 h before habitual bedtime, with an eating window of ~10 h/day on ≥6 days/week, adjusted to chronotype using stepwise phase-advance strategies where needed. Diet composition follows bariatric guidelines (protein, hydration, micronutrients). Timing logs and wearables track adherence; visits at 3, 6, and 12 months.
  Arms: Chronotype-Based Chrono-Nutrition (CB-CN)

SUMMARY:
This randomized controlled trial will evaluate the impact of chrono-nutrition, a dietary approach that aligns meal timing with the body's circadian rhythms, on weight change, metabolic outcomes, appetite, and gut microbiota in post-bariatric surgery patients. A total of 246 adults who underwent sleeve gastrectomy at least six months earlier will be enrolled at King Saud Medical City. Participants will be randomized to receive either standard post-bariatric nutritional care or personalized chrono-nutrition based on individual chronotype. Outcomes include weight change, metabolic biomarkers, dietary behaviors, sleep patterns, and gut microbiota composition. The study aims to determine whether integrating chrono-nutrition into post-bariatric follow-up can enhance metabolic health and improve long-term health.

DETAILED DESCRIPTION:
Bariatric surgery is the most effective treatment for severe obesity and often induces remission of comorbidities. However, up to 50-70% of patients experience weight recurrence and metabolic relapse within four years, suggesting that there must be adjunct strategies to sustain benefits. Circadian biology, the alignment of internal rhythms with behaviors such as eating and sleep, has emerged as a modifiable determinant of weight regulation, glycemic control, appetite, and inflammation. Chrononutrition, characterized by the deliberate scheduling of meals to correspond with circadian physiology, may present an innovative approach for long-term post-bariatric management. Early time-restricted eating (eTRE) has improved weight and metabolic outcomes in non-surgical populations. Post-bariatric patients may additionally benefit through improved hunger/satiety signaling, circadian alignment, favorable microbiota shifts, and possible epigenetic regulation. Despite this promise, randomized controlled evidence in post-bariatric cohorts is lacking.

Rationale and Significance This study addresses a major gap by evaluating whether chrononutrition tailored to chronotype improves long-term metabolic, microbial, and behavioral outcomes after bariatric surgery. Findings may reduce weight regain, enhance glycemic control, optimize gut microbiota composition, and offer information about circadian-epigenetic mechanisms. Results could inform future clinical practice guidelines and integrate precision nutrition into bariatric care.

Study Aim and Objectives The primary aim is to evaluate the effect of chronotype-based chrononutrition on metabolic, microbial, epigenetic, and behavioral outcomes in post-bariatric patients.

Primary Objective: Assess whether chronotype-based meal timing improves weight maintenance, insulin sensitivity, and gut microbiota diversity compared with standard care and generic eTRE.

Secondary Objectives: Examine effects on circadian gene expression, DNA methylation and histone modifications, gut hormones (GLP-1, PYY, ghrelin), eating behavior, sleep, mood, and physical activity. Explore microbiota and epigenetic mediation of outcomes.

Hypotheses Patients assigned to chrono-nutrition will demonstrate improved weight maintenance, metabolic outcomes, and circadian alignment compared to standard care. Chrononutrition is expected to alter gut microbiota favorably, epigenetic markers, and behavioral outcomes, with greater benefits observed when meal timing matches chronotype.

Study Design This is a randomized controlled trial at King Saud Medical City, Riyadh. Adult patients 6 months post-sleeve gastrectomy will be recruited from the bariatric nutrition clinic. Written informed consent is required.

Sample Size and Randomization

Based on power calculations, 246 participants (82 per group) will be randomized (1:1:1) to:

Control Group, standard post-bariatric care without meal timing.

eTRE Group, all meals consumed between 8:00 AM-6:00 PM.

Chronotype-Based Group: meal timing tailored to chronotype (morning, intermediate, evening).

Randomization will be stratified by chronotype. Follow-up visits will occur at baseline, 3, 6, and 12 months.

Inclusion Criteria Adults 18-65 years, ≥6 months post-sleeve gastrectomy, BMI 25-40 kg/m², ≥50% excess weight loss, cleared for a regular diet.

Exclusion Criteria:

Pregnancy, severe psychiatric illness, major unrelated chronic disease, revision bariatric surgery, prior intermittent fasting regimens, or use of medications affecting circadian rhythm.

Blinding:

Due to the nature of interventions, participants and dietitians cannot be blinded. Laboratory staff and statisticians will remain blinded to group allocation.

Assessments:

Anthropometry: weight, BMI, %EWL, waist circumference, bioimpedance body composition.

Biochemical markers: fasting glucose, insulin (HOMA-IR),HgbA1c, lipids, CRP, IL-6, TNF-α, leptin, adiponectin, ghrelin, GLP-1, PYY, cortisol, and vitamin D.

Gut microbiota: stool samples analyzed via 16S rRNA sequencing; SCFAs measured with GC-MS; bile acids via LC-MS.

Epigenetics: blood samples analyzed for DNA methylation (CLOCK, BMAL1, PER2, CRY1), histone modifications, and circadian gene expression (qRT-PCR).

Behavioral outcomes: validated questionnaires for sleep (PSQI), mood (BDI, GAD-7), and eating behavior (TFEQ, VAS appetite scores). Physical activity and sleep will also be objectively measured with actigraphy/wearable devices.

Dietary Habits: will be measured using Dietary Habit Questionnaire

Data Collection Timeline Baseline (6 months post-surgery), then follow-ups at 3, 6, and 12 months. Digital logs and wearable devices will track eating and activity behaviors continuously.

Statistical Analysis:

Primary outcomes will be analyzed with repeated-measures ANOVA and linear mixed models to compare groups over time. Microbiota diversity will be assessed using PERMANOVA and LEfSe analyses. Epigenetic and behavioral outcomes will be tested with ANCOVA and regression models. Mediation and moderation analyses (SEM) will explore pathways linking chrono-nutrition, microbiota, and metabolic outcomes. Intention-to-treat analysis will be performed, with multiple imputation for missing data.

Ethics The study follows the Declaration of Helsinki and is approved by the Ethics Committees of King Saud Medical City and King Saud University. Written informed consent is mandatory, and data will be anonymized.

Expected Impact:

This is the first RCT to test chronotype-based chrono-nutrition in post-bariatric patients. If effective, it could provide a scalable precision nutrition strategy to reduce weight regain, enhance metabolic outcomes, and guide future clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years who underwent Sleeve Gastrectomy (SG) 6 Months prior to enrollment.
* Have achieved ≥50% of excess weight loss post-surgery (to ensure initial success).
* Current BMI between 25-40 kg/m².
* No major postoperative complications and cleared for a regular diet by their healthcare provider.
* Participants must be able to align their eating schedule within a daytime window (morning to evening), ensuring that the first meal is consumed in the early part of the day and the last meal is completed before late evening, in accordance with chrono-nutrition guidelines.

Exclusion Criteria:

* • Pregnancy or planned pregnancy during the study period, and post menopaused females

  * Current diagnosis of severe psychiatric illness that may interfere with adherence (e.g., untreated major depression, psychosis, severe eating disorders).
  * Active malignancy or serious chronic disease unrelated to obesity that may confound outcomes (e.g., advanced renal failure, uncontrolled liver disease).
  * Use of medications known to significantly alter circadian rhythm or metabolism (e.g., corticosteroids, melatonin therapy) within the last 3 months.
  * Inability to comply with study requirements (dietary interventions, sample collection, or follow-up visits).Participants who have previously undergone revision bariatric surgery.
  * Individuals following intermittent fasting regimens prior to the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 246 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight maintenance and insulin sensitivity | Baseline, 3 months, 6 months, and 12 months
  Evaluate the effect of personalized chrono-nutrition interventions (early time-restricted eating and chronotype-based nutrition) on weight loss maintenance and insulin sensitivity in post-bariatric patients.

SECONDARY OUTCOMES:
Change in gut microbiota diversity and composition | Baseline, 6, 12 months
  Assess alpha/beta diversity, SCFA production, and bile acid profiles
Change in circadian gene expression and epigenetic markers | Baseline, 3, 6, 12 months
  DNA methylation (CLOCK, BMAL1, PER2, CRY1), histone modifications (H3Kac, H3K4me3, H3K27me3), and qRT-PCR expression (BMAL1, CLOCK, PPARα, GLUT4
Change in gut-derived hormones | Baseline and 12 months
  Fasting ghrelin, GLP-1, and PYY
Change in inflammatory markers and lipid profile | Baseline, 6, 12 months
  CRP, IL-6, TNF-α, total cholesterol, HDL, LDL, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Amani A Al-Farraj, Master, Principal Investigator — King Saud University
Locations (1):
- King Saud Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
ndividual participant data (IPD) will not be shared due to patient privacy concerns and institutional regulations.